CLINICAL TRIAL: NCT06881498
Title: A Substudy of the Effect of Acute Normovolemic Hemodilution in Bone Tumor Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024 0584
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Bone Tumor; Acute Normovolemic Hemodilution; Goal-Directed Fluid Therapy
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acute normovolemic hemodilution group (ANH group) (Experimental): The ANH process was initiated after tracheal intubation. After completion of ANH, goal-directed fluid therapy will begin until the end of the surgery.
  Interventions: Procedure: acute normovolemic hemodilution
- Standard Group (STD group) (No Intervention): After tracheal intubation, goal-directed fluid therapy will be implemented until the end of the surgery.

INTERVENTIONS:
Procedure: acute normovolemic hemodilution — The ANH was conducted with more than 8 ml/kg of whole blood drawn from an internal jugular introducer by gravity and collected into standard sterile blood storage bags containing citrate phosphate-dextrose anticoagulant. The allowable blood loss was capped according to the preoperative hemoglobin, estimated blood volume, and the target hemoglobin (10 g/dL). The collected blood was simultaneously replaced by an equal volume of succinyl gelatin solution via at least one large bore peripheralvenous catheter to maintain hemodynamic stability.
  Arms: acute normovolemic hemodilution group (ANH group)

SUMMARY:
The prevention of perioperative anemia has the potential to reduce complications, hospital stays, and long-term prognosis in patients undergoing bone tumor surgery. Data from previous studies suggest that the clinical efficacy of acute normovolemic hemodilution (ANH) has always been controversial, and intraoperative fluid administration strategy is an important confounding factor. The HEAL trial will assess whether ANH will improve postoperative hemoglobin levels when applying goal-directed fluid therapy in patients undergoing bone tumor surgery.

DETAILED DESCRIPTION:
Bone tumor surgery is associated with a significant risk of perioperative blood loss, with blood loss usually in the range of approximately 500-1000 ml. The postoperative anemia caused by blood loss is an independent risk factor for postoperative complications in patients undergoing bone tumor surgery, as well as affecting the long-term survival rate of cancer patients.

Acute normovolemic hemodilution (ANH) is a patient blood management measure. The clinical efficacy of acute normovolemic hemodilution (ANH) has always been controversial, and intraoperative fluid administration strategy is an important confounding factor. As goal-directed fluid therapy (GDFT) is increasingly used in clinical practice, it is of great importance to explore the efficacy of ANH in patients undergoing fluid management using GDFT.

Bone tumor surgery is an ideal setting to evaluate ANH in GDFT, as the procedure is associated with high blood loss and infusion. This trial has been designed as a randomized, controlled trial to determine whether ANH will improve postoperative hemoglobin levels when applying GDFT in patients undergoing bone tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 75 years;
2. undergoing elective bone tumor resection surgery;
3. preoperative hemoglobin ≥11 g/dL;

Exclusion Criteria:

1. using a tourniquet;
2. palliative operation or minimally invasive surgery;
3. BMI<18.5 or >30Kg/m^2;
4. international normalized ratio (INR) >1.5 or platelet count <100 × 10^9/L;
5. cardiopulmonary insufficiency;
6. hepatic and renal dysfunction;
7. active infectious disease;
8. allergy to succinyl gelatin;
9. pregnancy;
10. declined participation in the study or declined blood transfusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration on the first day after surgery | The first day after surgery
  The concentration of hemoglobin on the first day after surgery

SECONDARY OUTCOMES:
The rate of perioperative transfusion of allogeneic blood products | From the start of surgery to discharge or the 7th day following the operation, which comes first
  This includes blood products such as plasma and platelets, erythrocytes
The blood loss during the perioperative period | From the start of surgery to discharge or the 7th day following the operation, which comes first
  The volume of blood loss
The volume of fluid administration during the intraoperative period | From the beginning to the end of the surgery
  This includes intraoperative crystalloid infusion volume and intraoperative colliod infusion volume
The coagulation function tests during the perioperative period | From the start of surgery to discharge or the 7th day following the operation, which comes first
  This includes thromboelastography result
Perioperative embolic events | From the start of surgery to discharge or the 7th day following the operation, which comes first
  This includes thrombosis and embolism
Perioperative pulmonary infection | From the start of surgery to discharge or the 7th day following the operation, which comes first
  Diagnose according to radiologic examination, sign and symptom
Perioperative wound infection | From the start of surgery to discharge or the 7th day following the operation, which comes first
  Diagnose according to sign, symptom

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China